CLINICAL TRIAL: NCT00540956
Title: Descriptive Study Evaluating the Presence and Function of Natural Killer Cells in Elderly Patients With Acute Myeloid Leukemia in First Remission.
Brief Title: Natural Killer Cells in Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000564106; IPC-LAM-NK; INCA-RECF0429; IPC-2006/002
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2009-07

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Congenital Abnormalities | interventions — Cytarabine

INTERVENTIONS:
Drug: cytarabine
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying natural killer cells in samples of blood from patients with cancer may help doctors find out how these cells are effected by chemotherapy.

PURPOSE: This clinical trial is studying natural killer cells in older patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the evolution of functional receptors of natural killer (NK) cells after completion of chemotherapy in elderly patients with acute myeloid leukemia in first remission.

Secondary

* Measure the kinetics of cytotoxic functional recovery of NK cells.
* Determine activation markers of NK cells.

OUTLINE: This is a multicenter study.

Patients receive 1 course of consolidation therapy comprising an anthracycline and cytarabine to induce first remission.

Blood is collected on day 0 of the consolidation course and then every 2 weeks for 8 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia

  * No promyelocytic leukemia
  * No prior therapy

PATIENT CHARACTERISTICS:

* Hemoglobin > 10 g/dL

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-11; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Evolution of functional natural killer (NK) cells after chemotherapy

SECONDARY OUTCOMES:
Kinetics of NK cells
Activation markers of NK cells

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Vey, MD — Institut Paoli-Calmettes
Locations (1):
- Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille, France